CLINICAL TRIAL: NCT04594512
Title: Fresh Corneal Lenticule Implantation and Autologous Serum - New Approach in Treatment of Advanced Keratoconus Disease - Case Report
Brief Title: Fresh Corneal Lenticule Implantation and Autologous Serum - Case Report
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EyeHospitalP
Record Dates: First submitted 2020-10-01; First posted 2020-10-20 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Keratoconus; Keratoconus of Right Eye; Keratoconus, Unstable, Right Eye
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LENTICULE IMPLANTATION (Other): The present study may suggest that this procedure safely, reliably, and effectively increases corneal thickness and improves visual acuity with no adverse effects. It may even provide new avenues in the treatment of corneal ectasia. Stem cells and live keratocytes are well organized based on cornea transparency and in anterior segment OCT.
  Interventions: Other: Fresh corneal lenticule and autologous serum in advanced keratoconus using ReLex Smile surgery

INTERVENTIONS:
Other: Fresh corneal lenticule and autologous serum in advanced keratoconus using ReLex Smile surgery — A 19-year-old female patient with keratoconus and chronic hydrops cornea referred to the cornea department of our clinic with thin cornea and hydrops in chronic stage and minimal dry eye symptoms. Minimum corneal pachymetry in the right eye was 378 µm as measured by optical coherence tomography(AS-OCT-Zeiss). Atlas corneal topography showed steep K-values 82.60 ax.37 and flat K 75.15 D ax 127 with -7.45 corneal astigmatism. Her best corrected visual acuity was 0.0.5 in right eye and 1.0 in the left eye. Slit lamp examination showed intense punctate epitheliopathy (Figure 1), tear film break-up time (TBUT) was measured as 7-8 sec and Schirmer test was 10 mm in right eye, and the other eye examinations were determined normally
  Other Names: ReLex Smile

SUMMARY:
The aim of our study is to investigate the feasibility and the effect of fresh lenticule implantation as allogenic graft that will be taken from myopic patients to implant in patients with keratoconus disease using VisuMax Femtosescond laser- Smile module surgery with primary objective to increase central corneal thickness and secondary to improve visual acuity and reduces K-values and to show the autologous serum drop improve the recovery of patients with mild dry eye in keratoconus disease.

DETAILED DESCRIPTION:
A 19-year-old female patient with keratoconus and chronic hydrops cornea referred to the cornea department of our clinic with thin cornea and hydrops in chronic stage and minimal dry eye symptoms. Minimum corneal pachymetry in the right eye was 378 µm as measured by optical coherence tomography(AS-OCT-Zeiss). Atlas corneal topography showed steep K-values 82.60 ax.37 and flat K 75.15 D ax 127 with -7.45 corneal astigmatism. Her best corrected visual acuity was 0.0.5 in right eye and 1.0 in the left eye. Slit lamp examination showed intense punctate epitheliopathy (Figure 1), tear film break-up time (TBUT) was measured as 7-8 sec and Schirmer test was 10 mm in right eye, and the other eye examinations were determined normally.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age, male or female, of any race
* Willingness and ability to follow all instructions and comply with schedule for follow-up visits
* For females: Must not be pregnant

Exclusion Criteria:

* Contraindications, sensitivity or known allergy to the use of the test article(s) or their components
* If female, pregnant

Ages: 19 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Treatment of advanced keratoconus disease | 12 months
  Change of corneal central thickness using fresh lenticule with stromal stem cells, live keratocites and autologous serum

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT04594512/ICF_000.pdf